CLINICAL TRIAL: NCT07212868
Title: The Role of Glucagon in Glucose Metabolism in Humans With and Without Bariatric Surgery
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marzieh Salehi, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: STUDY00001597; R01DK141843 (NIH)
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Non-Diabetic
Keywords: glucagon; glucose metabolism; bariatric surgery

STUDY DESIGN:
Intervention Model Description: Placebo controlled physiologic study
Who Masked: Participant
Masking Description: Masking for participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mixed Meal study with and without glucagon receptor antagonist (Experimental): Mixed meal test conducted with a sequential design of receiving a single dose subcutaneous injection of glucagon receptor antagonist or placebo.
  Interventions: Drug: REMD-477 versus Placebo
- Pancreatic clamp (hypoglycemia and hyperglycemic) with and without glucagon infusion (Other): A cross-over study to compare the effect of glucagon infusion on glucose metabolism measured during clamp studies
  Interventions: Other: Exogenous glucagon versus saline infusion

INTERVENTIONS:
Drug: REMD-477 versus Placebo — Placebo versus glucagon receptor antagonist using a human monoclonal antibody with a high level of antagonistic effect against human glucagon receptor.
  Arms: Mixed Meal study with and without glucagon receptor antagonist
Other: Exogenous glucagon versus saline infusion — The effect of increased glucagon concentrations in plasma on glucose metabolism during glucose clamp will be studied.
  Arms: Pancreatic clamp (hypoglycemia and hyperglycemic) with and without glucagon infusion

SUMMARY:
The goal of this study is to understand the role of glucagon signal on glucose metabolism in individuals with and without bariatric surgery. The study is involved with measuring glucose metabolism with glucagon infusion and glucagon receptor blockade. We use an investigational drug called REMD 477. "Investigational" means that the has not yet been approved by the U.S. Food & Drug Administration (FDA). REMD-477 is a monoclonal antibody (an antibody made by cloning a unique white blood cell) that blocks the effect of glucagon.

DETAILED DESCRIPTION:
Participants will be screened, and if eligible will be enrolled for metabolic studies for two separate aims. In aim 1, they undergo glucose clamp study with and without glucagon infusion.

In aim 2, they undergo 2-day meal studies with and without a single dose administration of investigational drug, REMD 477 using a small needle subcutaneously. During these studies glycemic profile will be evaluated using CGM (Continuous glucose monitoring). Participants will also have a blood draw for liver enzymes8 weeks after the administration of REMD 477.

Participants will spend up to 3- 6 months participating in any pair study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form from participant.
2. Male or female, ≤65 and ≥18 years old
3. Subjects with history of gastric bypass surgery and sleeve gastrectomy more than a year since surgery and non-surgical subjects without history of gastrointestinal (GI) surgery
4. HbA1c ≤6%
5. Willing to adhere to the study intervention regimen
6. Female subjects of childbearing potential must have a negative pregnancy test at screening and all the study visits, and must not be lactating
7. Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception from screening and must agree to continue using such precautions during the study.It is strongly recommended for the male partner of a female subject to also use male condom plus spermicide throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

1. Diabetes
2. Pregnancy/lactation
3. Hgb <11
4. Current GI obstruction or chronic diarrhea
5. Subjects who are not within the age range of 18- 65 years.
6. Evidence of active cardiorespiratory, hepatic, gastrointestinal or renal disease.
7. History of allergy to the administered drugs.
8. History of, or any existing condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product, put the subject at risk, influence the subject's ability to participate or affect the interpretation of the results of the study and/or any subject unable or unwilling to follow study procedures.
9. Substance dependence or history of alcohol abuse and/or excess alcohol intake
10. Patients on ketogenic diet
11. Prisoners or institutionalized individuals
12. AST (SGOT) > 3 times upper limit of normal
13. ALT (SGPT) > 3 times upper limit of normal
14. History of clinical hypoglycemia documents based on Whipples' triad (ONLY for Aim 2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Glycemc response to meal ingestion | 0 to 240 minutes
  Changes in glucose response to meal ingestion occurred by administration of glucagon receptor antagonist (GRA).
Endogenous glucose production (EGP) during clamp studies | 0 to 240 minutes
  Changes in EGP (measured by tracer technique) with and without glucagon infusion

SECONDARY OUTCOMES:
Prandial glucose kinetics | Baseline to 240 minutes
  Glucose flux with and without GRA administration
Plasma GLP-1, GIP, insulin and glucagon concentrations | 0 to 240 minutes
  Changes in these outcomes following meal ingestion with and without GRA administration
Glucose clearance and insulin and glucagon concentrations during clamp studies | 0 to 240 minutes
  Outcomes with and without glucagon infusion

CONTACTS AND LOCATIONS:
Overall Officials: Marzieh Salehi, MD, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Texas Diabetes Institute - University Health System, San Antonio, Texas
  - University of Texas San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data summary results will be published in ClinicalTrials.gov as required by law and research findings will be published in a peer reviewed scientific journal.
Supporting Information: Study Protocol, SAP
Time Frame: At study end after analysis of data.